CLINICAL TRIAL: NCT02677051
Title: Sulforaphane in Autism: A Treatment Trial to Confirm Phenotypic Improvement With Sulforaphane Treatment in a New Jersey (NJ) Population of Individuals With Autism
Brief Title: Sulforaphane in a New Jersey (NJ) Population of Individuals With Autism
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rowan University (Other)
Responsible Party: Principal Investigator, Steven Buyske, Ph.D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro20120001884; CAUT15APL013 (Other Grant/Funding Number: NJ Governor's Council, Autism)
Record Dates: First submitted 2016-01-28; First posted 2016-02-09 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Autism; Autistic Disorder; Autism Spectrum Disorder; Autistic Behavior
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Child Development Disorders, Pervasive | interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): About 15 subjects will be randomized into this arm, receiving pills with an inactive placebo.
  Interventions: Drug: Placebo
- Sulforaphane (Experimental): About 30 subjects will be randomized into this arm, receiving pills with glucoraphanin rich broccoli seed powder containing active myrosinase resulting in sulforaphane once ingested Doses will be weight dependent with each pill resulting in ~ 50 µmol sulforaphane.
  Body weight Dose of sulforaphane 34 kg ~ 50 µmol 68 kg ~ 100 µmol 102 kg ~ 150 µmol
  Interventions: Drug: Sulforaphane

INTERVENTIONS:
Drug: Sulforaphane — Sulforaphane (1-isothiocyanato-4R- (methylsulfinyl)butane) is an isothiocyanate derived from the action of the plant enzyme myrosinase on glucosinolates including glucoraphanin and comes from consumption of many cruciferous vegetables.
  Other Names: Avmacol
  Arms: Sulforaphane
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is a double blind treatment trial that will test if sulforaphane improves core symptoms in autism. The investigators expect to see clinical improvement in some of these areas. Sulforaphanes come from eating certain vegetables such as broccoli. The investigators will be using a preparation that gives specific and reproducible amounts. The investigators will also test specific chemicals and genes needed for sulforaphane usage to try to understand differences in response.

DETAILED DESCRIPTION:
This study is a double blind randomized treatment trial that will test if sulforaphane improves core symptoms in autism. It is designed to try to replicate a previous trial (ClinicalTrials.gov Identifier NCT01474993) which reported that the isothiocyanate, sulforaphane treatment led to improvement by multiple metrics. Significant improvement was seen in behavior as measured by the Aberrant Behavioral Checklist (ABC) and by the Social Responsiveness Scale (SRS). In addition a significantly greater number of participants receiving sulforaphane had improvement in social interaction, abnormal behavior, and verbal communication as per the Clinical Global Impression (CGI). In addition The investigators will attempt to account for some variability in response to sulforaphane treatment by testing alleles of genes that are relevant in sulforaphane metabolism. The investigators will also measure glutathione levels, which are also important in sulforaphane metabolism and are in part regulated by sulforaphane..

Sulforaphane is the most potent naturally occurring inducer of mammalian cytoprotective enzymes known. Therapeutic potential is based at least in part on their ability to up-regulate genes responsible for alleviation of oxidative stress and to regulate both the immune system and the inflammatory response

40 Males with autistic disorder will be randomly selected to receive either sulforaphane or placebo. Seven visits are required by the subjects including enrollment ,screening, baseline, weeks 4, 10 and 18 and a follow up visit at seek 22.

ELIGIBILITY:
Inclusion Criteria:

* Autistic disorder diagnosis.
* Age between 13-30 years.
* Male gender.

Exclusion Criteria:

* Absence of a parent or legal guardian and consent,
* Those that can not or will not complete all visits and adherence to study regimen.
* Seizure within 2 years of screening,
* Impaired renal function (serum creatinine> 1.2 mg/dl).
* Impaired hepatic function (> 2x upper limit of normal).
* Impaired thyroid function (TSH outside normal limits).
* Current infection or treatment with antibiotics.
* Chronic medical disorder (e.g., cardiovascular disease, stroke or diabetes) or major surgery within 3 months prior to enrollment.
* Less than 13 years or more than 30 years of age.
* Female gender.
* A diagnosis of autism spectrum disorder other than autistic disorder, for example, Asperger, Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS) etc.

Ages: 13 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2016-02; Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Aberrant Behavior Checklist (ABC) scores. | Baseline, week 4, week 10, week 18 and week 22.
Change in Social Responsiveness Scale (SRS) scores. | Baseline, week 4, week 10, week 18 and week 22.
Clinical Global Impression Severity Scale (CGI-S). | Baseline
Clinical Global Impression Improvement Scale (CGI-I) to measure change from baseline CGI-S scores. | Week 4, week 10, week 18 and week 22.

SECONDARY OUTCOMES:
Liver Function Tests as a screen for entry into the study and a monitor of potential change/adverse events due to treatment. | Baseline, week 4, week 18 and week 22.
Renal Function Tests as a screen for entry into the study and a monitor of potential change/adverse events due to treatment. | Baseline, week 4, week 18 and week 22.
Thyroid Stimulating Hormone (TSH) as a screen for entry into the study and a monitor of potential change/adverse events due to treatment. | Baseline, week 4, week 18 and week 22.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Buyske, Principal Investigator — Rutgers, The State University of NJ
Locations (1):
- Rutgers University - Staged Research Building, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh K, Connors SL, Macklin EA, Smith KD, Fahey JW, Talalay P, Zimmerman AW. Sulforaphane treatment of autism spectrum disorder (ASD). Proc Natl Acad Sci U S A. 2014 Oct 28;111(43):15550-5. doi: 10.1073/pnas.1416940111. Epub 2014 Oct 13. PMID 25313065

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT02677051/Prot_SAP_002.pdf
  • Informed Consent Form (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT02677051/ICF_003.pdf